CLINICAL TRIAL: NCT00466323
Title: The Effectiveness of FMPO in Improving the Quality of Care for Persons With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Maryland, Baltimore County (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 04-255; H-28791 (Other: UMB IRB)
Record Dates: First submitted 2007-04-24; First posted 2007-04-27 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Major Depression
Keywords: Mental Illness; Schizophrenia; Education; Family member treatment; Active psychoses
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Depressive Disorder, Major; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FMPO Condition (Experimental): Family Member Provider Outreach is a brief recovery oriented model. THe FMPO meets with the consumer for 2-3 sessions and with the family for 2-3 sessions with the consumer's permission.
  Interventions: Behavioral: Family Member Provider Outreach
- Enhanced treatment as usual (e-TAU) (Active Comparator): Enhanced treatment as usual. In this condition, the consumer is given a list of family services available including the family intervention team.
  Interventions: Behavioral: Enhanced treatment as usual (e-TAU)

INTERVENTIONS:
Behavioral: Family Member Provider Outreach — Family Member Provider Outreach is a brief recovery oriented model. THe FMPO meets with the consumer for 2-3 sessions and with the family for 2-3 sessions with the consumer's permission.
  Arms: FMPO Condition
Behavioral: Enhanced treatment as usual (e-TAU) — Enhanced treatment as usual. In this condition, the consumer is given a list of family services available including the family intervention team.
  Arms: Enhanced treatment as usual (e-TAU)

SUMMARY:
The purpose of this study is to learn how to help veterans play a stronger role in shaping their mental health care. Specifically we want to see if we can help veterans improve their mental health treatment by helping them decide if they want to involve family in their mental health treatment, and if so, how. The study will compare a "family member provider" program to an "enhanced treatment as usual approach" in achieving these goals.

DETAILED DESCRIPTION:
Previous research demonstrates that when families are active participants in the clinical care of persons with SMI, veterans experience improved outcomes, including treatment retention, vocational services participation, and empowerment. Numerous controlled trials show that when family involvement achieves the level of intensity and family psychoeducation (FPE), relapse rates are cut in half, and treatment adherence, clinical symptoms, and patient functioning are improved. However, despite these demonstrated benefits, rates of family involvement in the VA are unacceptably low. Even minimal family-clinician contact occurs for only one third of VA SMI patients, a lower rate than in non-VA systems of care. Therefore, it is not surprising that FPE, an intensive form of family-clinician contact, is almost never offered in the VA. In fact, a national VA survey conducted within the last three years indicated that 0% of VAs offer FPE programs conforming to EBP guidelines. Our previous experience further suggests that these deficits in care are due to combinations of provider, patient, and family factors, and that the VA presents specific challenges to implementing existing model programs, including FPE. We therefore believe it is necessary to approach the challenge of increasing family involvement in a step-wise fashion, first by engaging families in the processes of care, before trying to enlist them in more intensive programs such as FPE. Further, family engagement would likely be most effective if it builds on a foundation that empowers consumers to make informed choices regarding the involvement of relatives in care. Our group has developed and piloted a new, family-engagement approach that is gradual, patient-centered, recovery-based, and can address various barriers to improving care. It is manualized and thus replicable. The proposed study will implement and further evaluate this intervention, the brief Family Member Provider Outreach (FMPO).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Diagnosis of a psychotic disorder in keeping with criteria established by the Serious Mental Illness Treatment Research and Evaluation Center (SMITREC){{646}} (schizophrenic disorders (295.0-295.9), affective psychoses (296.1, 296.4-296.8) and other psychotic diagnoses (297.0-298.9)) or diagnosis of Major Depression with psychotic features (296.xx)
* Decisional capacity to provide informed consent
* At least two outpatient visits within last six months
* At least monthly face-to-face contact for one hour or more with a patient-identified family member or caregiver
* Assessment by the treating therapist or psychiatrist that the patient is clinically stable enough to participate in the program.

Family Member/Caregiver Inclusion Criteria

* Age 18-80 years
* Decisional capacity to provide informed consent
* Permission from veteran to be contacted

Exclusion Criteria:

* Patients whose families have attended the FPE group within the last six months
* Patients whose families have had at least monthly clinician contact in the last six months
* Patients who are currently homeless
* Patients who participated in the FMPO pilot.

Family Member/Caregiver Exclusion Criteria:

* Individuals who do not meet the inclusion criteria
* Individuals who participated in the FMPO pilot.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2007-09; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa B Dixon, MD MPH, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (2):
- United States (2):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland

REFERENCES:
- [Result] Glynn SM, Dixon LB, Cohen A, Murray-Swank A. The Family Member Provider Outreach program. Psychiatr Serv. 2008 Aug;59(8):934. doi: 10.1176/ps.2008.59.8.934. No abstract available. PMID 18678695
- [Result] Cohen AN, Drapalski AL, Glynn SM, Medoff D, Fang LJ, Dixon LB. Preferences for family involvement in care among consumers with serious mental illness. Psychiatr Serv. 2013 Mar 1;64(3):257-63. doi: 10.1176/appi.ps.201200176. PMID 23242515
- [Result] Dixon LB, Glynn SM, Cohen AN, Drapalski AL, Medoff D, Fang LJ, Potts W, Gioia D. Outcomes of a brief program, REORDER, to promote consumer recovery and family involvement in care. Psychiatr Serv. 2014 Jan 1;65(1):116-20. doi: 10.1176/appi.ps.201300074. PMID 24177229

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We enrolled (consented and baseline) 238 individuals. Over the course of the study, we withdrew 6 individuals. We only conducted analysis on the 232 remaining individuals.
Period: Overall Study
Arm/Group | FMPO Condition | Enhanced Treatment as Usual (e-TAU)
Started | 117 | 115
Completed | 89 | 92
Not Completed | 28 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMPO Condition | Enhanced Treatment as Usual (e-TAU) | Total
Number analyzed (Participants) | 117 | 115 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (9.4) | 51.2 (8.7) | 51.5 (9.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 114 | 109 | 223
  >=65 years | 3 | 6 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 97 | 98 | 195
Region of Enrollment [Number; unit: participants]
  United States | 117 | 115 | 232

OUTCOME MEASURES:

1. Primary Outcome: Family-Clinician Contact (Including Contact With FMPO Clinician)
Description: Chart review looking at the any clinician contact with veteran's family members
Time Frame: Within 6 months of intervention
Population: We enrolled (consented and baseline) 238 individuals. Over the course of the study, we withdrew 6 individuals. We only conducted analysis on the 232 remaining individuals.
Measure: Mean (Standard Deviation); unit: Number of Interactions
Arm/Group | FMPO Condition | Enhanced Treatment as Usual (e-TAU)
Number analyzed (Participants) | 111 | 115
Number of Interactions
  Pre Test (Baseline) | .4 (2.0) | .3 (.9)
  Post Test (Within 6 months of the intervention) | 1.6 (2.3) | .3 (1.0)

2. Secondary Outcome: Consumer's Recovery Rating - MHRM Total Score
Description: We measured recovery attitudes and beliefs with the Mental Health Recovery Measure (MHRM), a 30-item self-report measure that has a total score and eight subscales.The MHRM scales range from 0-120, with a higher score indicating better recovery.
Time Frame: Within 6 months of intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | FMPO Condition | Enhanced Treatment as Usual (e-TAU)
Number analyzed (Participants) | 111 | 115
Units on a Scale
  Pre Test (Baseline) | 75.6 (17.3) | 77.0 (19.1)
  Post Test (Within 6 months of the intervention) | 80.2 (18.7) | 79.9 (20.4)

3. Secondary Outcome: Consumer's Recovery Rating - MHRM - Overcoming Stuckness Sub Score
Description: We measured recovery attitudes and beliefs with the Mental Health Recovery Measure (MHRM), a 30-item self-report measure that has a total score and eight subscales. This sub score is Overcoming Stuckness.The MHRM sub scales range from 0-16, with a higher score indicating better recovery.
Time Frame: Within 6 month of the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FMPO Condition | Enhanced Treatment as Usual (e-TAU)
Number analyzed (Participants) | 111 | 115
units on a scale
  Pre Test (Baseline) | 10.6 (2.5) | 11.4 (2.5)
  Post Test (Within 6 months of the intervention) | 11.4 (2.6) | 11.3 (2.3)

4. Primary Outcome: Family-Clinician Contact (Not Including Notes From FMPO Clinicians)
Description: Chart review looking at the any clinician contact with veteran's family members
Time Frame: Within 6 months of intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Interactions
Arm/Group | FMPO Condition | Enhanced Treatment as Usual (e-TAU)
Number analyzed (Participants) | 111 | 115
Number of Interactions
  Pre Test (Baseline) | .4 (2.0) | .3 (.9)
  Post Test (Within 6 months of the intervention) | .5 (2.0) | .3 (1.0)

ADVERSE EVENTS:
Arm/Group | FMPO Condition | Enhanced Treatment as Usual (e-TAU)
Serious Adverse Events (participants affected / at risk) | 2/117 | 1/115
Other Adverse Events (participants affected / at risk) | 0/117 | 0/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMPO Condition (N=117) | Enhanced Treatment as Usual (e-TAU) (N=115)
Hospitalization (Psychiatric disorders) | 2 (2) | 1 (1) — Psychiatric hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes